CLINICAL TRIAL: NCT04312399
Title: Hormone Replacement Trial Against ALzheimers' Disease
Acronym: HARALD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EC/2018/0315
Record Dates: First submitted 2020-01-08; First posted 2020-03-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Postmenopausal Symptoms; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: 10 study groups: 9 groups who start with hormonal treatment and 1 control group who doesn't start with hormonal treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- oral hormonal therapy (Other): Postmenopausal women who start with oral hormonal therapy (Progesteron + uterogestan) according to standard of care practice. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- transdermal hormonal therapy (Other): Postmenopausal women who start with transdermal hormonal (Oestrogel + uterogestan) therapy according to standard of care practice. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- oral hormonal therapy + hysterectomy (Other): Postmenopausal women who start with oral hormonal therapy (progesteron) according to standard of care practice and had a hysterectomy in the past. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- transdermal hormonal therapy + hysterectomy (Other): Postmenopausal women who start with transdermal hormonal therapy (Oestrogel ) according to standard of care practice and had a hysterectomy in the past. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- oral hormonal therapy + IUD (Other): Postmenopausal women who start with oral hormonal therapy (Progynova) according to standard of care practice and have already an intra-uterine device. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- transdermal hormonal therapy + IUD (Other): Postmenopausal women who start with transdermal hormonal therapy (Oestrogel ) according to standard of care practice and have an intra-uterine device. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- selective oestrogenreceptor modulators (Other): Postmenopausal women who start with hormonal therapy according to standard of care practice and take selective oestrogenreceptor modulators (Nolvadex) because of their cancer in their medical history. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- aromatase inhibitors (Other): Postmenopausal women who start with hormonal therapy according to standard of care practice and who taken aromatase inhibitors (Femara) because of their cancer in their medical history. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- Duavive (Other): Postmenopausal women who start with hormonal therapy according to standard of care practice and who take duavive because of their cancer in their medical history. Before the start of the treatment blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take
- Control (Other): Postmenopausal women who don't start with hormonal therapy according to standard of care practice. At the first study visit blood will be taken and 6 (and 12) months after the start of the therapy blood will be taken for analysis. At the 2/3 study visits the patient will be asked to complete the questionaires (TANGO-SF, ICIQ, Cohen, Pittsburgh sleep quality). Only at the first study visit an MMSE test will be taken, to make sure the patient has no dementia.
  Interventions: Procedure: blood take

INTERVENTIONS:
Procedure: blood take — Blood is taken to analyse degradation products of the metabolism of amyloid

SUMMARY:
The influence of postmenopausal hormone treatment on dementia is not clear. Dysfunctions in the metabolism of amyloid in the disease of Alzheimer result in an elevated presence of degradation products in cerebrospinal fluid.

The degradation products in blood will be analysed during the trial, to get better insight in menopause and the start of hormonal therapy.

Postmenopausal women with and without history of breast cancer will be recruited for the trial.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* 40 - 65 years

Exclusion Criteria:

* Longer than 10 years in menopause
* thyroid dysfunction
* hypertension
* medical history of psychiatric comorbidity
* Alcohol and/or drug abuse
* medical history of neurologic symptoms with cognitive symptoms

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Degradation products of the Amyloid metabolism in blood | 2 years after the first patient was included, the first batch of samples will be analysed.
  The influence of hormone treatment (menopause) and anti-hormone treatment (breastcancer) on the amyloid metabolism and the development of Alzheimer will be evaluated. Different laboratory analysis will be performed to evaluate the degradation products of the metabolism of amyloid in blood. Different parts of the degradation products will be analysed namely: Plasma total-tau
Degradation products of the Amyloid metabolism in blood | 2 years after the first patient was included, the first batch of samples will be analysed.
  The influence of hormone treatment (menopause) and anti-hormone treatment (breastcancer) on the amyloid metabolism and the development of Alzheimer will be evaluated. Different laboratory analysis will be performed to evaluate the degradation products of the metabolism of amyloid in blood. Different parts of the degradation products will be analysed namely: Nurofilament light chain
Degradation products of the Amyloid metabolism in blood | 2 years after the first patient was included, the first batch of samples will be analysed.
  The influence of hormone treatment (menopause) and anti-hormone treatment (breastcancer) on the amyloid metabolism and the development of Alzheimer will be evaluated. Different laboratory analysis will be performed to evaluate the degradation products of the metabolism of amyloid in blood. Different parts of the degradation products will be analysed namely: Abeta1-40
Degradation products of the Amyloid metabolism in blood | 2 years after the first patient was included, the first batch of samples will be analysed.
  The influence of hormone treatment (menopause) and anti-hormone treatment (breastcancer) on the amyloid metabolism and the development of Alzheimer will be evaluated. Different laboratory analysis will be performed to evaluate the degradation products of the metabolism of amyloid in blood. Different parts of the degradation products will be analysed namely: Abeta1-42
Degradation products of the Amyloid metabolism in blood | 2 years after the first patient was included, the first batch of samples will be analysed.
  The influence of hormone treatment (menopause) and anti-hormone treatment (breastcancer) on the amyloid metabolism and the development of Alzheimer will be evaluated. Different laboratory analysis will be performed to evaluate the degradation products of the metabolism of amyloid in blood. Different parts of the degradation products will be analysed namely: YKL-40
Degradation products of the Amyloid metabolism in blood | 2 years after the first patient was included, the first batch of samples will be analysed.
  The influence of hormone treatment (menopause) and anti-hormone treatment (breastcancer) on the amyloid metabolism and the development of Alzheimer will be evaluated. Different laboratory analysis will be performed to evaluate the degradation products of the metabolism of amyloid in blood. Different parts of the degradation products will be analysed namely: Neurogranin
APOE-genotyping in blood | 2 years after the first patient was included, the first batch of samples will be analysed.
  The influence of hormone treatment (menopause) and anti-hormone treatment (breastcancer) on the amyloid metabolism and the development of Alzheimer will be evaluated. APOE-genotyping will be performed
identify BACE1 in blood | 2 years after the first patient was included, the first batch of samples will be analysed.
  The influence of hormone treatment (menopause) and anti-hormone treatment (breastcancer) on the amyloid metabolism and the development of Alzheimer will be evaluated. BACE1 will also be identified in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Depypere, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent university hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided